CLINICAL TRIAL: NCT04349046
Title: Exception Cementless Femoral Stem in Total Hip Arthroplasty. A Multicenter, Retrospective and Prospective, Non-controlled Post Market Clinical Follow-up Study (Implants and Instrumentation)
Brief Title: Exception Cementless Hip Stem
Acronym: Exception
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2018-45H
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis, Hip; Rheumatoid Arthritis; Inflammatory Arthritis; Congenital Hip Dysplasia; Avascular Necrosis of Hip; Femoral Neck Fractures
Keywords: Total hip arthroplasty; Medical device; Performance; Safety; Hip prosthesis; Clinical benefits
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Arthritis; Hip Dislocation, Congenital; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patient who received the Exception stem: Patient who received the Exception stem between January 2008 and September 2012 and consented to the original data collection.
  Interventions: Device: Total hip arthoplasty (THA)

INTERVENTIONS:
Device: Total hip arthoplasty (THA) — Total hip arthroplasty (THA) is a common operative treatment where an arthritic, degenerative or fractured hip joint is replaced with a prosthetic device if conservative options are unable to relieve pain and debilitating symptoms. THA was traditionally performed on patients over 60 years old, but now includes young and active patients, as well as very old ones thanks to the continuous improvement in implant design. Major indications of THA include osteoarthritis, rheumatoid arthritis, avascular necrosis and hip fractures. The THA surgical procedure involves replacing the head of the femur and acetabulum or socket with an artificial prosthesis. This system is composed of a femoral stem that is inserted into the femoral canal, a ball that attaches to the femoral stem, and an acetabular component or shell that replaces the acetabulum.

SUMMARY:
This study is a multicenter, retrospective and prospective, non-controlled, non-randomized post market clinical follow-up study. The objectives of this study are to confirm the long-term safety, performance and clinical benefits the Exception Cementless femoral stem (standard and varized) when used in primary total hip arthroplasty.

DETAILED DESCRIPTION:
Six surgeons have prospectively collected clinical data for patients operated consecutively between January 2008 and September 2012. The patients have been operated based on the indications and contraindications listed in the Instructions For Use (IFUs) of the implant.

This study is an extension of the surgeons' data collection as an attempt from Zimmer-Biomet to fulfill its post-market surveillance obligations by recovering clinical data retrospectively and prospectively.

Study Procedure Flowchart - retrospective data collection: most patients had clinical follow-ups at pre-op, operative, immediate post-op, 3 Months, 1 year, 2, 3, 5, 7 years post-surgery during which their surgeons collected clinical data. This data will therefore only be collected by Zimmer-Biomet after the patients specifically consent to it.

Study Procedure Flowchart - prospective data collection: The informed consent signed by the patient for this study also allow Zimmer Biomet to collect the data of the standard clinical follow-up that will be conducted by the investigators at least 10 years post-surgery.

ELIGIBILITY:
At the time of surgery, the inclusion criteria were based on the indications presented in the IFUs:

* Primary or secondary osteoarthritis
* Inflammatory impairment of the hip, rheumatoid arthritis, etc.
* Fracture of the neck of the femur
* Avascular necrosis of the femoral head
* Sequelae from previous operations on the hip, osteotomies, etc.
* Congenital hip dysplasia.
* Patient is older than 18 years old
* Patient had consented to the original data collection after his/her surgery

At the time of surgery, the exclusion criteria were based on the contraindications presented in the IFUs:

* Local or systemic infections.
* Serious muscular, neurological or vascular deficiencies in the limb concerned.
* Bone destruction or poor quality bone likely to affect the stability of the implant (Paget's disease, osteoporosis, etc.)
* Any concomitant disorder likely to affect the function of the implant.
* Allergy to one of the implant components.
* Patients weighing more than 110 kg.
* Patient incapable of following the recommendations of the surgeon

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Six surgeons have prospectively collected clinical data for patients operated consecutively between January 2008 and September 2012. The patients have been operated based on the indications and contraindications listed in the Instructions For Use (IFUs) of the implant.
  For this retrospective and prospective study, only the patients who had consented to the original data collection after their surgery will be contacted.
  These the patients should be capable of understanding the surgeon's explanations and following his instructions, should be able and willing to participate in the last follow-up visit, and should give consent to take part in the study. The patients should meet all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Implant survival based on removal or intended removal of the device and determined using the Kaplan-Meier method | 10 years post-surgery

SECONDARY OUTCOMES:
Pain and functional performance based on the Harris Hip Score | 10 years post-surgery
  The score is given from 0 to 100 with Excellent: 90 - 100, Good: 80 - 89, Fair: 70 - 79, and Poor: < 70
Subject quality-of-life determined by the EQ-5D (EuroQoI) score | 10 years post-surgery
  The lowest score (0) corresponds to "the worst health the patient can imagine", and the highest rate (100) corresponds to "the best health he can imagine".
X-rays evaluated for radiolucencies, osteolysis, hypertrophy, subsidence, heterotopic ossification, etc | 10 years post-surgery
Safety based on eventual complications occurred including dislocations and revisions/removals | 10 years post-surgery]

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (6):
- Hôpital Princesse Paola, Aye, Belgium
- France (5):
  - CH Alpes Léman, Contamine-sur-Arve
  - CH Annecy Genevois, Épagny
  - Hopital Renee Sabran, Hyères
  - Clinique Basseres Kacem-Boudhar, Nîmes
  - Hôpitaux Du Léman, Thonon-les-Bains

IPD SHARING:
Plan to Share IPD: No